CLINICAL TRIAL: NCT02574221
Title: A Pilot Study to Evaluate the Sensitivity of a Novel Molecular Method for Plaque Toxicity
Brief Title: A Pilot Study to Evaluate a Molecular Method for Plaque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2015049
Record Dates: First submitted 2015-10-09; First posted 2015-10-12 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Plaque; Gingivitis
MeSH Terms: conditions — Plaque, Amyloid; Gingivitis | interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stannous fluoride toothpaste (Experimental): brush twice a day for 8 weeks
  Interventions: Drug: stannous fluoride toothpaste
- cavity protection toothpaste (Sham Comparator): brush twice a day for 8 weeks
  Interventions: Drug: cavity protection toothpaste

INTERVENTIONS:
Drug: stannous fluoride toothpaste — 0.454% stannous fluoride toothpaste
  Arms: stannous fluoride toothpaste
Drug: cavity protection toothpaste — 0.243% sodium fluoride toothpaste
  Arms: cavity protection toothpaste

SUMMARY:
This study is to evaluate the sensitivity of the molecular method and its ability to split a stannous fluoride toothpaste versus a negative control.

ELIGIBILITY:
Inclusion Criteria:

In order to be included in the study, each subject must:

* Provide written informed consent to participate in the study;
* Be 18 years of age or older;
* Agree not to participate in any other oral/dental product studies during the course of this study;
* Agree to delay any elective dentistry (including dental prophylaxis) until the study has been completed;
* Agree to maintain their current oral hygiene routine between the Screening and Baseline Visit and not to add/change their oral care products during this time;
* Agree to refrain from any form of non-specified oral hygiene during the treatment periods (after the Baseline Visit), including but not limited to the use of products such as floss or whitening products;
* Agree to return for all scheduled visits and follow study procedures;
* Must have at least 16 natural teeth;
* Be in good general health, as determined by the Investigator/designee based on a review of the health history/update for participation in the study;
* Agree to refrain from all oral hygiene for at least 12 hours prior to each visit;
* Agree to refrain from eating, chewing gum, drinking and using tobacco for 4 hours prior to each visit;
* Have at least 20 bleeding sites (sites with a score of 1 or 2 on the GBI index);
* Have minimum 3 sampling sites with bleeding and pocket depth ≥3mm but not deeper than 4mm;
* Have minimum 3 sampling sites without bleeding and with pocket depth ≤2mm.

Exclusion Criteria:

Subjects are excluded from study participation where there is evidence of:

* Have had a dental prophylaxis within 2 weeks of plaque sampling visits;
* Have taken antibiotics or used anti-gingivitis / anti-bacterial oral care products such as chlorhexidine or Listerine within 2 weeks of plaque sampling visits;
* Have rampant caries, open or untreated caries, or advanced periodontitis requiring prompt treatment;
* Need an antibiotic prophylaxis prior to dental visits;
* A history of hypersensitivity to oral care products containing stannous fluoride;
* A history of hypersensitivity to dyes (from products containing food dyes);
* Present with any disease or condition(s) that could be expected to interfere with examination procedures or the subject's safe completion of the study; or
* Are pregnant (Self-reported) or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
plaque scores | baseline
plaque scores | week 8

SECONDARY OUTCOMES:
gingivitis score | baseline
gingivitis score | week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States